CLINICAL TRIAL: NCT03057405
Title: Intra-operative (IO) Navigation and IO-CBCT for 3D Orbital Reconstruction in Post-traumatic and Post-ablative Defects. Evaluation of the Potential of a Fully Integrated Brainlab Iplan System.
Brief Title: Intra-operative (IO) Navigation and IO-CBCT for 3D Orbital Reconstruction
Status: Completed | Type: Observational
Sponsor: AZ Sint-Jan AV (Other)
Responsible Party: Principal Investigator, Johan Abeloos, head of department, AZ Sint-Jan AV
Other Study IDs: B049201731057
Record Dates: First submitted 2017-02-10; First posted 2017-02-20 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Orbital Fractures
Keywords: intra-operative navigation; 3D virtual planning; intra-operative cone beam computed tomography (CBCT)
MeSH Terms: conditions — Orbital Fractures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- intra-operative CBCT
- 3D virtual planning + intra-operative navigation
- 3D virtual planning + intraoperative navigation + IO CBCT

SUMMARY:
Background Correction of post traumatic and post-ablative orbita defects remains a challenge for the maxillofacial surgeon. The purpose of such intervention is the restoration of both function and aesthetics by anatomical reconstruction of the bony orbitawalls, with attention to the orbitavolume. Unfortunately, the results of such interventions today are still somewhat unpredictable.

The aim of this study is to determine whether 3D virtual planning combined with intra-operative navigation can increase the predictability of the outcome in function and aesthetics.

Study design Retrospective study. Demographic data, diagnostic and surgical parameters will be collected of all patients undergoing orbital surgery between 01/01/2012 and 31/12/2016 at the department. Pre- en postoperative orbit volume will be determined based on CT-analysis in Brainlab software, and compared to the non-defected orbit.

ELIGIBILITY:
inclusion criteria

* patients of all genders
* patients of all ages
* patients undergoing surgery for orbit fractures between 01/01/2012 until 31/12/2016

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients undergoing surgery for orbit fractures between 01/01/2012 until 31/12/2016
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-01-10 (Actual)

PRIMARY OUTCOMES:
accuracy of orbital volume reconstruction, as measured in Brainlab | immediate postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Johan Abeloos, Principal Investigator — head of department

IPD SHARING:
Plan to Share IPD: No